CLINICAL TRIAL: NCT07264322
Title: Observational Imaging Study on Real-Time Dynamic Changes of Normal Pharyngolaryngeal Structures During Barium Swallow in Patients Undergoing Routine Barium Meal Examination
Brief Title: Real-Time Dynamic Imaging Study of Normal Pharyngolaryngeal Structures During Barium Swallow (GLAM-III)
Acronym: GLAM-III
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Jiangling, Principal Investigator, Zhejiang Cancer Hospital
Other Study IDs: IRB-2025-1096（IIT）
Record Dates: First submitted 2025-09-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Barium Meal Examination
Keywords: Barium Swallow; Pharyngolaryngeal Dynamic Changes; Pyriform Sinus; Cricoid Cartilage Lamina; Laryngeal Mask Design

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The integrity and functional stability of pharyngolaryngeal anatomical structures are critical for airway management, and the dynamic changes of key structures (e.g., pyriform sinus, cricoid cartilage lamina) during swallowing directly relate to the design and clinical safety of laryngeal masks. This observational study aims to investigate the real-time dynamic changes and physiological movement patterns of normal pharyngolaryngeal structures during barium swallow using routine barium meal examination imaging. The findings will provide anatomical and physiological evidence for optimizing laryngeal mask design and improving its anatomical fit with the pharynx and larynx.

DETAILED DESCRIPTION:
After approval by the Ethics Committee of Zhejiang Cancer Hospital (Approval Number: IRB-2025-1096(IIT)), this study will be registered on ClinicalTrials.gov prior to participant enrollment. Given that the study only utilizes de-identified imaging data from routine barium meal examinations (no additional procedures or interventions for participants), informed consent is exempted as approved by the Ethics Committee. The study is planned to be conducted from August 2025 to October 2025.

Eligible participants are patients undergoing routine barium meal examinations at Zhejiang Cancer Hospital, meeting the inclusion criteria (18-75 years old, no pharyngolaryngeal surgery/trauma/congenital malformation, no swallowing dysfunction, unobstructed oropharyngeal-esophageal pathway, etc.) and excluding those with contraindications (e.g., goiter compressing pharyngolaryngeal structures, barium allergy).

Barium Swallow Examination Procedure:

All procedures follow the standard clinical protocol for barium meal examinations, with no additional radiation exposure or burden on participants:

Static Imaging (Resting State): Participants assume a standing position. A digital X-ray machine (Shimadzu Uni-vision) is used to obtain static images of the pharyngolaryngeal region, recording the baseline anatomical positions of the pyriform sinus, cricoid cartilage lamina, and esophageal inlet.

Dynamic Imaging (Swallowing State): Participants are instructed to swallow 5ml, 10ml, 20ml, and 40ml of medical barium sulfate suspension (concentration: 160-200% W/V) sequentially. During swallowing, a dynamic fluoroscopic imaging system is activated (frame rate: 15 frames/second) to continuously record the entire process of barium passing from the oropharynx through the larynx to the esophagus (each swallowing event lasts approximately 5-10 seconds). Each participant repeats the swallowing action 4-5 times, and the clearest dynamic image sequence is selected for subsequent analysis.

Data Collection and Analysis:

Image analysis software is used for frame-by-frame parsing of dynamic images. Key anatomical structures (pyriform sinus boundaries, anterior edge of the cricoid cartilage lamina, esophageal inlet center) are labeled, and coordinate positioning technology is applied to analyze the following parameters:

Displacement and angle changes of pharyngolaryngeal structures from resting state to peak swallowing phase; Preferred pathway of barium through the oropharynx (unilateral pyriform sinus, bilateral pyriform sinuses, or central region of the cricoid cartilage lamina); Retention time of barium in the pyriform sinus and its passing speed; Expansion amplitude of the pyriform sinus and displacement distance of the cricoid cartilage lamina during swallowing

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* No history of pharyngolaryngeal surgery, trauma, or congenital malformation;
* No swallowing dysfunction, pharyngolaryngeal inflammation, or neurological diseases affecting swallowing;
* No recent use of drugs that affect muscle function (e.g., muscle relaxants, anticholinergics);
* Barium meal examination confirms unobstructed oropharyngeal-esophageal pathway;
* Normal pharyngolaryngeal anatomical structure (confirmed by preliminary imaging review);
* Scheduled to undergo routine barium meal examination at Zhejiang Cancer Hospital for clinical diagnosis.

Exclusion Criteria:

* Presence of diseases that may compress pharyngolaryngeal structures (e.g., goiter, mediastinal mass);
* Allergy to barium sulfate or other components of the barium suspension.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient scheduled to take barium meal examination
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Real-time dynamic changes of pharyngolaryngeal structures during swallowing | From the initiation of the barium swallow to the complete passage of the bolus through the upper esophageal sphincter, as assessed under videofluoroscopy (an average of 15 minutes per participant).
  Measurement of displacement distance of the cricoid cartilage lamina, expansion amplitude of the pyriform sinus, and movement trajectory of the esophageal inlet during swallowing (assessed via dynamic fluoroscopic imaging).

SECONDARY OUTCOMES:
Proportion of participants with consistent instrument insertion pathway and barium's preferred pathway (pyriform sinus) | From the initiation of the barium swallow to the complete passage of the bolus through the upper esophageal sphincter, as assessed under videofluoroscopy (an average of 15 minutes per participant).
  Analysis of the consistency between the barium's preferred pathway (pyriform sinus) and the insertion pathway of laryngeal mask-related instruments, to explain the anatomical fit differences among three laryngeal mask designs (LMA Supreme, I-gel, GMA-Tulip).

OTHER OUTCOMES:
Barium flow speed through the oropharynx | From the initiation of the barium swallow to the complete passage of the bolus through the upper esophageal sphincter, as assessed under videofluoroscopy (an average of 15 minutes per participant).
  The speed of barium flow through the oropharyngeal region, measured by videofluoroscopic swallowing study. The speed will be calculated by tracking the movement of the barium bolus head between two predefined anatomical points (e.g., the pyriform sinus and the lower edge of the cricoid cartilage) and reported in millimeters per second (mm/s)
Preferred pathway of barium flow | From the initiation of the barium swallow to the complete passage of the bolus through the upper esophageal sphincter, as assessed under videofluoroscopy (an average of 15 minutes per participant).
  The primary anatomical pathway of the barium bolus as it passes the laryngeal inlet, assessed by videofluoroscopy. The pathway will be categorized as either passing through the pyriform sinuses or through other channels (e.g., directly over the arytenoids). The result will be reported as the proportion (percentage) of participants with barium flow primarily through the pyriform sinuses.
Displacement of the cricoid cartilage lamina during barium swallow | From the initiation of the barium swallow to the complete passage of the bolus through the upper esophageal sphincter, as assessed under videofluoroscopy (an average of 15 minutes per participant).
  The extent of posterior-inferior displacement of the cricoid cartilage lamina during the pharyngeal phase of swallowing, measured on lateral videofluoroscopic images. The displacement will be quantified as the vertical distance (in millimeters) from the resting position of the cricoid cartilage to its maximum displaced position.

CONTACTS AND LOCATIONS:
Overall Officials: Pingbo Xu, Ph. D, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Jiangling Wang, Hangzhou, Zhejiang, China